CLINICAL TRIAL: NCT03334071
Title: Exercise regiMens Before and duRing Advanced Cancer thErapy: A Pilot Study to Investigate Improvements in Physical Fitness With Exercise Training Programme Before and During Chemotherapy in Advanced Lung Cancer Patients.
Brief Title: Exercise Intervention During Chemotherapy in Advanced Lung Cancer Patients
Acronym: EMBRACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RHM CAN 0960; 13/YH/0354 (Other: Research Ethics Committee)
Record Dates: First submitted 2017-10-26; First posted 2017-11-07 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Non Small Cell Lung Cancer; Non Small Cell Lung Cancer Stage IIIB; Non Small Cell Lung Cancer Metastatic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Exercise intervention
Who Masked: Investigator, Outcomes Assessor
Masking Description: Cardiopulmonary exercise testing assessor, outcome/toxicity assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise Intervention (Active Comparator): Patients in the intervention arm will participate in a supervised in-hospital, exercise training program on a cycle ergometer before and during chemotherapy. At week 5-6 there will be a transition period of in-hospital to home-based exercise training (at this point we will perform the exercises that they will perform at home in the in-hospital environment to ensure that the patient understands the home-based exercise training programme) and then week 7-12 will be home-based exercise training only with telephone support.
  Interventions: Behavioral: Exercise
- Negative Control (No Intervention): Patients in the control arm will not undergo an exercise training program.
- Observational (No Intervention): Patients who do not enrol in RCT will be enrolled in the observational arm

INTERVENTIONS:
Behavioral: Exercise — High intensity interspersed with short periods of exercise at a moderate intensity (aerobic interval training). We will also include resistance training in each session.
  The supervised in-hospital exercise training sessions will last <1 hour, exercise training intensities will be individually tailored to each CPET. Exercise training will involve repeated exercise bouts of 3 minutes at a moderate exercise intensity (80%AT) followed by 2 minutes of exercise at a high intensity (50%Δ) for a predetermined amount of time.
  The home-based training programme will involve stair climbing (where possible) and brisk walking to achieve heart rates commensurate with those achieved during the in-hospital exercise training sessions.
  Arms: Exercise Intervention

SUMMARY:
Trial Phase: Pilot

Indication: Stage IIIB/IV NSCLC

Primary Objective: To assess the feasibility and tolerability of exercise training during palliative chemotherapy.

Secondary Objective: 1) To assess fitness levels in patients undergoing palliative chemotherapy, and to explore whether exercise training can prevent a reduction in fitness.

2) To determine the baseline fitness, as assessed by cardiopulmonary exercise testing (CPET), of a cohort of patients with stage IIIb/IV non small cell lung cancer who are about to initiate treatment with chemotherapy 3) To compare patients enrolled in the EMBRACE randomized controlled trial (RCT) with those who decline.

4)To investigate any relationship between baseline fitness and outcomes including therapy related complications, response, and survival in those patients who decline exercise training or are randomized to observation.

5) To assess the feasibility of the translation of in-hospital exercise training to home-based training during chemotherapy.

6) To document the effects of chemotherapy on cellular energetics and mitochondrial function.

Rationale: Chemotherapy has a detrimental effect on physical fitness, and this effect can be later reversed by training. The investigators wish to understand the mechanism of this detrimental effect, and investigate whether it can be prevented or attenuated by giving chemotherapy concurrently with exercise training.

Trial Design: Randomised controlled study (1:1) comparing chemotherapy alone, with chemotherapy plus exercise training. A subgroup of patients will have muscle biopsies. Patients who decline randomisation will be offered enrolment into an observational arm.

Sample size : 100 patients (to include 48 who will be randomised, and 52 in the observational arm).

DETAILED DESCRIPTION:
EMBRACE is a multi-centre pilot study for 100 patients with EGFR negative NSCLC undergoing first line platinum based chemotherapy. It is a prospective randomised (1:1) 2-arm controlled study. A nested mechanism study will be performed in a sub group of patients willing to have muscle biopsies.

Patients will be randomised to the exercise intervention or the control arm. All patients will undergo standard chemotherapy with gemcitabine and carboplatin (or equivalent) for 12 weeks. Patients randomised to the intervention arm will undergo concurrent exercise training during their 12 weeks of chemotherapy treatment. Patients randomised to the control arm will undergo chemotherapy only. During the 12 weeks of the study, assessments will be performed on all patients (including CPET tests and HRQL questionnaires). The exercise training sessions and study assessments will not affect timing of delivery of chemotherapy. Patients who decline randomisation will be offered entry into an observational study.

The follow-up phase will commence when patients have completed 12 weeks of chemotherapy, or sooner for patients who stop chemotherapy early due to progressive disease or toxicity. During the follow-up phase data will be for survival and to follow any AEs related to study procedures. AEs not related to study procedures will not require follow up. Ongoing chemotherapy after week 12 will be as per investigator and patient choice, and may include further induction cycles, maintenance chemotherapy, or observation.

In a subgroup of willing patients muscle biopsies will be performed at baseline, during chemotherapy, and after completion of chemotherapy.

TRIAL OUTCOME MEASURES

The primary outcome variables for this feasibility and tolerability study will be adherence to the exercise training program, and adverse events.

The secondary outcome variables will be response to chemotherapy, fitness levels as measured by Cardiopulmonary Exercise Testing (CPET), Time to get up and go test (TUG), grip strength, bioimpedance, CT measures of cancer cachexia, and Montreal score, cancer related symptoms, HRQL, and activity levels.

The exploratory outcome variables will be overall survival, toxicity, and biomarkers of stress and cellular energetics.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged over 18 years old
* Histologically or cytologically confirmed NSCLC (adenocarcinoma, squamous cell carcinoma, large cell carcinoma, undifferentiated carcinoma or other)
* Stage IIIb/IV disease
* Patients being treated with first line gemcitabine and platinum based chemotherapy (other equivalent regimens may be considered on discussion with Judith Cave)
* Performance status 0-2 (PS 2 have to be deemed fit enough to complete all cycles of chemotherapy).

Exclusion Criteria:

* Unable to consent
* Under 18 years
* Unable to perform CPET
* Significant cardiac ischaemia of > 1.5mm symptomatic and > 2mm asymptomatic observed on the baseline ECG
* Weight of >145kg (weight limit for cycle ergometer)
* Any other contraindication to CPET based on ACCP/ATS Guidelines and summarised in the table below.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-04-04 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants completing exercise sessions as a function of the whole programme. | 12 weeks
  Adherence to the exercise training program
Adverse events | 12 weeks
  Common Terminology on Complications (CTC AE v4)

SECONDARY OUTCOMES:
Fitness levels as measured by Cardiopulmonary exercise testing (CPET) | 12 weeks
  Physical fitness - oxygen uptake at anaerobic threshold
Timed up and go test (TUG) | 12 weeks
  Physical fitness
Grip strength | 12 weeks
  Physical fitness
Montreal score - Prognostic survival score | 12 weeks
  Non small cell lung cancer stage, CRP, albumin, lactic acid dehydrogenase (LDH) and absolute neutrophil count/lymphocyte count ratio (N/L).
Health related quality of life questionnaire | 12 weeks
  FACT-L quality of life questionnaire
Health related quality of life questionnaire | 12 weeks
  Dukes Activity Status Index
Health related quality of life questionnaire | 12 weeks
  International Physical Activity Questionnaire (IPAQ)
Health related quality of life questionnaire | 12 weeks
  Godin Leisure Time Questionnaire (GLTEQ).
Physical activity | 12 weeks
  Patients will wear a Sensewear Pro3 activity monitor (armband) or similar e.g. AX3 3-Axis Logging Accelerometer (wristband) for 72 hours. Number of steps in a 72 hours period will be calculated
Survival | 1 year
  Overall survival
Response to chemotherapy | 12 weeks
  Cross sectional imaging will be performed within 12 days of the third cycle of chemotherapy, to assess response to treatment. Scans will be reported according to the Response Evaluation Criteria for Solid Tumours (RECIST Version 1 http://www.irrecist.com/recist/recist-in-practice/01.html).
Fitness levels as measured by Cardiopulmonary exercise testing (CPET) | 12 weeks
  Physical fitness - oxygen uptake at peak exercise

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Jack, PhD, Principal Investigator — University Hospitals Southampton NHS Foundation Trust
Locations (1):
- University Hospitals Southampton NHS Foundation Trust, Southampton, United Kingdom